CLINICAL TRIAL: NCT01144572
Title: A Prospective, Multicenter, Non-interventional Study to Evaluate Quality of Life in Chinese Postmenopausal HR(+) EBC Patients During Adjuvant Aromatase Inhibitors(AIs) Treatment
Brief Title: Quality of Life in Chinese Postmenopausal HR(+) Early Breast Cancer (EBC) Patients During Adjuvant Aromatase Inhibitors(AIs) Treatment
Acronym: BC Qol NIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OCN-ARI-2010/1
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: Quality of Life; postmenopausal HR(+); Early Breast Cancer; adjuvant AI treatment; Quality of Life in Chinese postmenopausal HR(+) EBC patients during adjuvant Aromatase Inhibitors(AIs) treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Chinese postmenopausal HR(+) EBC patients during adjuvant Aromatase Inhibitors(AIs) treatment

SUMMARY:
The purpose of the study is to evaluate quality of life (Qol) in postmenopausal HR (+) EBC patients during adjuvant AIs treatment in terms of: the change of the trial outcome index (TOI) of the FACT-B questionnaire from baseline to 24 months. This study will recruit approximately 500 patients from 21 sites in China. The patients should be postmenopausal HR (+) EBC patients who have already start adjuvant AIs treatment but within 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women ≤ 70 years old, with histologically proven HR (+) early breast cancer.
* Undergoing upfront AIs adjuvant treatment within 7 days.

Exclusion Criteria:

* Patients who disagree to participate this study
* Patients who, for whatever reason (eg, confusion, infirmity), are unlikely to comply with trial requirements.
* The AIs have not been approved by SFDA for the indication of upfront adjuvant endocrine therapy in early breast cancer.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible patients will be recruited when they start their upfront AIs adjuvant treatment within 7 days.
Sampling Method: Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The change of the trial outcome index (TOI) of the FACT-B questionnaire from baseline to 24 months. | 24 months

SECONDARY OUTCOMES:
The change of the trial outcome index (TOI) of the FACT-B questionnaire from baseline to 6 months, 12 months and 18 months | 6-18 months
The change of the emotional well-being (EWB) subscales score of the FACT-B questionnaire from baseline to 6 months, 12 months, 18 months and 24 months | 6-18 months
The change of the social well-being (SWB) subscales score of the FACT-B questionnaire from baseline to 6 months, 12 months, 18 months and 24 months. | 6-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Shao Zhimin, Principal Investigator — Fudan University; Karen Atkin, Study Director — AstraZeneca; Xu Johnson, Study Chair — AstraZeneca
Locations (15):
- China (15):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Guiyang, Guizhou
  - Research Site, Harbin, Heilongjiang
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Ningbo, Zhejiang
  - Research Site, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Cao A, Zhang J, Liu X, Wu W, Liu Y, Fan Z, Zhang A, Zhou T, Fu P, Wang S, Ouyang Q, Tang J, Jiang H, Zhang X, Pang D, He J, Shi L, Wang X, Sheng Y, Mao D, Shao Z. Health-related quality of life of postmenopausal Chinese women with hormone receptor-positive early breast cancer during treatment with adjuvant aromatase inhibitors: a prospective, multicenter, non-interventional study. Health Qual Life Outcomes. 2016 Mar 24;14:51. doi: 10.1186/s12955-016-0446-2. PMID 27009092